CLINICAL TRIAL: NCT04918550
Title: A Survey on the Cognition and Use of Intraosseous Access Among Emergency Medical Staff
Brief Title: A Survey on the Cognition and Use of Intraosseous Access Among Medical Staff
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0396
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Intraosseous Access

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no drug and device — there is no intervention

SUMMARY:
A Survey on the Cognition and Use of Intraosseous Access among Emergency Medical Staff, which is based on the platform of "WJX.CN", from January 5, 2018 to January 23, 2018, via local emergency-related academic organizations to emergency medical staff throughout the country. There are 3 sections in the questionnaire: the demographic information of the participants; cognition levels and clinical use of IO; barriers and attitudes towards clinical use of IO including willingness, confidence and training demand.

DETAILED DESCRIPTION:
This research is a cross-sectional survey research, using the method of network survey, with domestic emergency medicine medical staff as the research object. Inclusion criteria: 1) Emergency medical staff who have a Chinese medical practitioner certificate or a nurse practitioner certificate and are within the valid registration period; 2) Agree to participate in this study. Exclusion criteria: incomplete questionnaires. The questionnaire was designed for the "Survey of Current Status of Marrow Cavity Pathway Cognition of Medical Staff in Emergency Department", including three parts: (1) general information of the survey object; (2) cognition and use status of IO; (3) clinical application of IO Attitude. Based on the "Questionnaire Star" platform, questionnaires are distributed through various emergency-related academic organizations. The front page of the questionnaire clearly marked the reminder of voluntary participation in the survey and related declarations, and it could be filled out after informed consent.

ELIGIBILITY:
Inclusion Criteria: 1) Emergency medical staff who have a Chinese medical practitioner certificate or a nurse practitioner certificate and are within the valid registration period; 2) Agree to participate in this study.

Exclusion Criteria: incomplete questionnaires.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical staff of emergency medicine in china
Sampling Method: Non-Probability Sample
Enrollment: 3194 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Cognition levels and clinical use of IO | two weeks
  Cognitive level is divided into: never heard of, heard of, equipped, used

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency Medicine, Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No
no share